CLINICAL TRIAL: NCT03535012
Title: Sensory Recovery of Reconstructed Breast With Breast Reconstructive Options
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1019
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of 5 mm3 including skin tissue from the flap for reconstruction at the time of immediate breast reconstruction A sample of 5 mm3 including skin tissue at the time of nipple reconstruction (nipple reconstruction will be performed at the time requested by the subject)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reconstruction using an implant: Immediate 2 stage implant based breast reconstruction after mastectomy. All expanders are placed in the subpectoralis muscle using ADM as a sling. After expansion of the tissue expander change to the permanent implant is performed.
- Reconstruction using abdominal tissue: immediate free DIEP flap breast reconstruction after mastectomy. DIEP(deep inferior epigastric perforator) free flap was prepared and transferred to the breast pocket. Microanastomosis was done under the microscopic magnification. On sitting position, free flap was inset into breast pocket with confirming of satisfactory inflammatory fold.

SUMMARY:
Over the past 10 years, there have been substantial improvements in breast reconstruction by plastic surgeons, and much has been achieved in aesthetic restoration after mastectomy. Advances in both microsurgery and implants have allowed for a wider variety of surgical methods, and procedural skills that minimize donor site complications have been developed.

With such satisfactory aesthetic results, interest has recently increased not only in breast reconstruction but also in sensory recovery. Due to the growing expectation of patients, sensory discomfort may decrease overall patient satisfaction with breast reconstruction despite good aesthetic results. Hence, for qualitative improvement of breast reconstruction surgery, efforts must be made to restore sensation in the reconstructed breast. There has been little research on the mechanism of sensory recovery despite its clinical importance. This study aimed to compare the degree of sensory recovery in the reconstructed breast using various reconstruction methods as well as to evaluate the status of neural regeneration with harvesting the tissues when nipple reconstruction is performed.

ELIGIBILITY:
Inclusion Criteria:

* Female adults over 20 years of age
* Patients who have undergone or plan to undergo total mastectomy and immediate breast reconstruction after the diagnosis of breast cancer (including carcinoma in situ)
* written consent to study participation

Exclusion Criteria:

* presence of neuropathy that may hinder accurate assessment of sensation
* presence of dermatological condition that may hinder accurate assessment of sensation
* inability to provide written consent
* decided by the research team to be unsuitable for this study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted by dividing the subjects into two groups(25 per each arm) according to the method of reconstruction: implant vs. abdominal tissue. It is difficult to determine a sample size that can establish statistical significance based on previous studies. Therefore, the number of targeted subjects was estimated based on the number of patients that can generally be recruited during the study period.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Sensory recovery in the reconstructed breast according to reconstructive options | 3 months (±1 month) after immediate breast reconstruction surgery
  Subjects will be followed up with quantitative sensory testing at 3 months (±1 month) after immediate breast reconstruction surgery.
Sensory recovery in the reconstructed breast according to reconstructive options | 6 months (±1 month) after immediate breast reconstruction surgery
  Subjects will be followed up with quantitative sensory testing at 6 months (±1 month) after immediate breast reconstruction surgery.
Sensory recovery in the reconstructed breast according to reconstructive options | 12 months (±2 months) after immediate breast reconstruction surgery
  Subjects will be followed up with quantitative sensory testing at 12 months (±2 months) after immediate breast reconstruction surgery.
Sensory recovery in the reconstructed breast according to reconstructive options | 18 months (±2 months) after immediate breast reconstruction surgery
  Subjects will be followed up with quantitative sensory testing at 18 months (±2 months) after immediate breast reconstruction surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic Surgery, Yonsei University School of Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No